CLINICAL TRIAL: NCT05597748
Title: Modified Herbst Approach to Improve Chin Projection in Class II Malocclusion Patients: A Randomized Controlled Trial
Brief Title: Modified Herbst Approach to Improve Chin Projection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00124682
Record Dates: First submitted 2022-10-11; First posted 2022-10-28 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Class II Malocclusion
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Intervention Model Description: Four parallel arms all under treatment
Who Masked: Outcomes Assessor
Masking Description: The patient and care provider can't be masked as it is obvious what appliance modification is being used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Class II type A malocclusion - proclination of upper incisors indicated - No TADs (Active Comparator): A hybrid Herbst appliance approach will be used (current available conventional treatment). The upper jaw component will be a maxillary expander secured on the first molar bands. The lower arch would have an uncemented lower acrylic full-coverage splint-type. In between Herbst-type pistons will be used. Upper brackets will be initially bonded and upper incisors proclined until normal inclination values are attained.
  Interventions: Device: Conventional Herbst Approach
- Class II type B malocclusion - proclination of upper incisors not indicated - No TADs (Active Comparator): A hybrid Herbst appliance approach will be used (current available conventional treatment). The upper jaw component will be a maxillary expander secured on the first molar bands. The lower arch would have an uncemented lower acrylic full-coverage splint-type. In between Herbst-type pistons will be used.
  Interventions: Device: Conventional Herbst Approach
- Class II type A malocclusion - proclination of upper incisors indicated - TADs (Experimental): A modified hybrid Herbst appliance approach (same hybrid Herbst appliance approach but with the addition of temporary anchorage devices (TADs) in both arches) will be used (alternative treatment). In the upper arch, the TADs would be inserted in the paramedical palatal area. In the lower arch, they would be inserted buccally between the roots of the lower second premolar and the first permanent molar. Elastomeric chains will be used to link these TADs to the first molars in the upper arch and to a buccal bottom on the lower canines. Upper brackets will be initially bonded and upper incisors proclined until normal inclination values are attained.
  Interventions: Device: Modified Herbst Approach
- Class II type B malocclusion - proclination of upper incisors not indicated - TADs (Experimental): CA modified hybrid Herbst appliance approach (same hybrid Herbst appliance approach but with the addition of temporary anchorage devices (TADs) in both arches) will be used (alternative treatment). In the upper arch, the TADs would be inserted in the paramedical palatal area. In the lower arch, they would be inserted buccally between the roots of the lower second premolar and the first permanent molar. Elastomeric chains will be used to link these TADs to the first molars in the upper arch and to a buccal bottom on the lower canines.
  Interventions: Device: Modified Herbst Approach

INTERVENTIONS:
Device: Modified Herbst Approach — A modified hybrid Herbst appliance approach (same hybrid Herbst appliance approach but with the addition of temporary anchorage devices (TADs) in both arches) will be used (alternative treatment). In the upper arch, the TADs would be inserted in the paramedical palatal area. In the lower arch, they would be inserted buccally between the roots of the lower second premolar and the first permanent molar. Elastomeric chains will be used to link these TADs to the first molars in the upper arch and to a buccal bottom on the lower canines. Upper brackets will be initially bonded and upper incisors proclined until normal inclination values are attained.
  Arms: Class II type A malocclusion - proclination of upper incisors indicated - TADs; Class II type B malocclusion - proclination of upper incisors not indicated - TADs
Device: Conventional Herbst Approach — A hybrid Herbst appliance approach will be used (current available conventional treatment). The upper jaw component will be a maxillary expander secured on the first molar bands. The lower arch would have an uncemented lower acrylic full-coverage splint-type. In between Herbst-type pistons will be used.
  Arms: Class II type A malocclusion - proclination of upper incisors indicated - No TADs; Class II type B malocclusion - proclination of upper incisors not indicated - No TADs

SUMMARY:
This study will collect data to try to assess which one of the two management options works better. The first option involves the use of the bite corrector first and then braces, while the second option involves the temporary addition of small support bone screws with the bite corrector later and then braces. Currently, it is not clearly known if there are important differences between the proposed management options. Such approaches are conventionally used in orthodontic practices. The information collected in this study will be used to compare the differences in the nature of the facial, teeth, and bone changes after the treatment. Questions about the experience while using the devices will be asked.

DETAILED DESCRIPTION:
Purpose

The present study will compare facial, skeletal, and dental changes among adolescents with mild to moderate Class II malocclusion using two Class II orthopedic orthodontic approaches. Patient-reported outcomes will also be assessed through validated questionnaires and qualitative interviews.

Hypothesis

Participants that use the modified Herbst approach do not showcase facial, dental, and skeletal changes that are different than those using the conventional Herbst approach.

Justification

One of the most common causes of a Class II malocclusion is a deficient mandibular projection (either due to reduced size or retruded position). Although in adults the only reasonable way to improve the mandibular projection is through surgical repositioning, in growing individuals an orthopedic alternative may significantly reduce the perceived need for this type of surgery later in life.

Several craniofacial orthopedic appliances have been used to attempt an orthopedic correction of Class II malocclusion of a mandibular origin, aiming to possibly improve functional, muscular, skeletal, and dental disharmonies.1,2,3 A wide array of related publications exist that have been summarized through several systematic reviews with or without meta-analysis.

The Herbst appliance is widely known for its relative effectiveness in correcting Class II malocclusions. It is most commonly used as a fixed appliance that repositions the jaw to a more anterior and downward position displacing the condyles away from the articular eminence.4,-8 This is thought to facilitate condylar bone apposition; hence, increasing mandibular size dimensions. Several papers have considered the efficiency of the Herbst appliance in Class II correction during early permanent dentition. But only one study evaluated changes produced by the Herbst appliance in mixed dentition patients and it concluded that the effects of the Herbst appliance were mainly dentoalveolar.5 Several different designs of the Herbst appliance have been reported in the literature.6-11

A modified Herbst approach by Manni has shown promising results. An increment in the mandibular chin projection of 5 mm has been reported. Due to the fact that the reported positive changes are so far only based on case reports and retrospective data12-24, a randomized controlled trial seems to be the next prudent step.

Objectives

Assess if the modified Herbst approach produces facial, dental, and skeletal changes that are different than those using the conventional Herbst approach.

Assess if the use of the modified Herbst approach facilitates a treatment experience (overall quality of life, oral health-related quality of life, and described experience) that is different than the one with the conventional Herbst approach.

Methods

Each potential participant will undergo an orthodontic clinical screening to determine if they fill the inclusion criteria (mild to moderate Class II malocclusion in a growing individual - two distinct Class II malocclusion phenotypes - see eligibility criteria below). Eligible individuals will be approached with an opportunity to participate in the research study. After understanding the research purpose and possible side effects, and if they choose to participate, they will voluntarily sign the informed consent form.

They will be randomly assigned to one of two groups. The allocation sequence will be done through randomization tables by a statistician and sealed envelopes generated. Once a willing participant is deemed to have fulfilled the inclusion criteria and provided informed consent the randomization will occur. For each Class II malocclusion type, two groups will be randomly generated.

Group 1 - Class II type A malocclusion - proclination of upper incisors indicated. A hybrid Herbst appliance approach will be used (current available conventional treatment). The upper jaw component will be a maxillary expander secured on the first molar bands. The lower arch would have an uncemented lower acrylic full coverage splint-type. In between Herbst-type pistons will be used. For Type, A upper brackets will be initially bonded and upper incisors proclined until normal inclination values are attained.

Group 2 - Class II type B malocclusion - proclination of upper incisors not indicated. A modified hybrid Herbst appliance approach (same hybrid Herbst appliance approach but with the addition of temporary anchorage devices (TADs) in both arches) will be used (alternative treatment). In the upper arch, the TADs would be inserted in the paramedical palatal area. In the lower arch, they would be inserted buccally between the roots of the lower second premolar and the first permanent molar. Elastomeric chains will be used to link these TADs to the first molars in the upper arch and to a buccal bottom on the lower canines. For Type, A initially upper brackets will be initially bonded and upper incisors proclined until normal inclination values are attained.

Both treatment arms will start as soon as the randomization has been done. Full orthodontic records (2D x-rays, photos, and dental casts) will be obtained for both groups at baseline and after this treatment phase is completed. Further comprehensive treatment will be offered to these patients as this initial management approach is not expected to fully align and level the teeth. This would be an additional elective option at an additional cost.

Two validated quality-of-life tools will be used. The CPQ11-14 assesses oral health-related quality of life and the EuroQoL assesses the overall quality of life. These two tools will be collected before and after this management approach. Additionally, a qualitative approach will be used at the end of the trial participants to better understand the participant's journey through the process.

Sample size

A sample of 40 patients (8 patients per treatment group are needed but the total sample is set to 10 considering a 20% loss during follow-up) will be sought. This sample was based on alfa of 5% and a beta of 20%. A clinically significant difference of 4.9 mm in Pg to OLp and a variance of 12.25 was set as clinically meaningful based on the pilot retrospective study by Manni et al.16.

n=f(a,b)*2SD2/Dif2 25

f(a,b)=7.85 (Table XIII page 22) 25

sd=12.25 Manni et al.16

Expected difference= 4.9 mm Pg to OLp Manni et al.16

ELIGIBILITY:
Inclusion Criteria:

* Class II skeletal malocclusion based on PgOLp more than 85 mm and A-OLp more than 75 mm.
* Perceived potential improvement of facial convexity.
* At least end-to-end bilateral molar relationship.
* Early permanent dentition.
* No congenitally missing teeth.

Exclusion criteria:

* Class II skeletal malocclusion based on PgOLp less than 85 mm and A-OLp less than 75 mm.
* Only reasonable management option is surgery.
* Less than an end-to-end bilateral molar relationship.
* Mixed dentition dentition.
* Congenitally missing teeth.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Skeletal chin prominence | 1 year
  Assess if the modified Herbst approach produces a more prominent chin protrusion than the one produced by the conventional Herbst. The distance in mm between the skeletal chin and a perpendicular virtual reference line will be calculated.
Lower incisor inclination | 1 year
  Assess if the modified Herbst approach produces less incisor inclination than the conventional Herbst approach. The angulation in degrees between the lower incisor and the mandibular plane will be calculated.
Overall quality of life | 1 year
  Assess if the overall quality of life is different than the one with the conventional Herbst approach. The CPQ11-14 ISF questionnaire will be used to assess oral health-related quality of life. The range of possible values es between 0 and 32. Lower values implied better perceived QoL.
Oral health-related quality of life | 1 year
  Assess if the oral health-related quality of life is different than the one with the conventional Herbst approach. The EuroQoL questionnaire will be used to assess oral health-related quality of life. The index calculates a value between 0 and 1. A higher value implies better QoL.
Soft tissue Chin prominence | 1 year
  Assess if the modified Herbst approach produces a more prominent chin protrusion. The distance in mm between the lower lip and a perpendicular virtual reference line will be calculated

SECONDARY OUTCOMES:
Maxillary lip prominence | 1 year
  Assess if the modified Herbst approach produces a less prominent lip protrusion. The distance in mm between the upper lip and a perpendicular virtual reference line will be calculated.
Mandibular lip prominence | 1 year
  Assess if the modified Herbst approach produces a more prominent lip protrusion. The distance in mm between the lower lip and a perpendicular virtual reference line will be calculated.
Upper incisor inclination | 1 year
  Assess if the modified Herbst approach produces less incisor inclination than the conventional Herbst approach. The angulation in degrees between the upper incisor and the maxillary plane will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Flores Mir, DSc, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Only the participant's unique ID is stored as personal identifying information. To be able to link this ID to specific participant identifiable information access to our password-protected health database would be needed.